CLINICAL TRIAL: NCT06268990
Title: Metabolic Outcome of Obese Subjects Receiving Fecal Microbiota Transplantation of Lean Versus Gastric Bypass Treated Subjects. A Pilot Study
Brief Title: FMT in Obesity: RYGB vs. LEAN vs. Autologous FMT
Acronym: DACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wiebke Kristin Fenske (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Sponsor-Investigator, Wiebke Kristin Fenske, Prof. Dr., University Hospital Bergmannsheil Bochum
Organization: University Hospital Bergmannsheil Bochum (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FE 1159/6-1
Record Dates: First submitted 2024-01-29; First posted 2024-02-21 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Morbid Obesity; Metabolic Syndrome; Diabetes; PreDiabetes; Insulin Resistance
Keywords: Fecal microbiota transfer; obesity; glucose homeostasis; bariatric surgery; gut microbiome
MeSH Terms: conditions — Obesity, Morbid; Metabolic Syndrome; Diabetes Mellitus; Prediabetic State; Insulin Resistance; Obesity | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RYGB-FMT intervention group (Active Comparator): morbidly obese patients randomized for FMT from patients successfully treated with RYGB surgery
  Interventions: Procedure: Fecal microbiota transplantation
- LEAN-FMT intervention group (Active Comparator): morbidly obese patients randomized for FMT from normal weight (lean) volonteers
  Interventions: Procedure: Fecal microbiota transplantation
- M-FMT intervention group (Sham Comparator): morbidly obese patients randomized for autologous FMT
  Interventions: Procedure: Fecal microbiota transplantation

INTERVENTIONS:
Procedure: Fecal microbiota transplantation — FMT is the transfer of fecal material containing gut microorganisms from a donor into the intestinal tract of a recipient
  Other Names: FMT

SUMMARY:
This double-blinded proof-of-concept study is proposed to explore the effects of fecal microbiota transfer (FMT) in human subjects. Here we perform FMTs into obese recipients using stool from lean unoperated donors and from previously obese patients after successfull treatment with bariatric Roux-en-Y Gastric Bypass (RYGB) surgery. Obese patients treated with their own material (autologous FMT) serve as controls. After FMT treatment the functional impact of post-surgery microbiome changes on host energy consumption and regulation of blood glucose levels will be analysed. Additionally the variations on the microbiota and metabolite composition will be profiled using extensive sequencing analyses. The major aim of the study is to explore the scientific rationale for targeted gut microbiota modulation in management of obesity and related metabolic diseases.We estimate the transfer of microbiota from RYGB donors is superior to the transfer of lean microbiota at inducing reduced adiposity and improving high blood glucose levels in obese recipients. Each is better than a sham procedure (autologous FMT), which itself can also induce considerable short-term effects.

DETAILED DESCRIPTION:
Patients and stool donors (for RYGB-/Lean-FMT-intervention groups) will be recruited at the Endocrinology outpatient clinic at the University Hospital of Graz. Patients will be randomized in a 1:1:1 manner. In all three study groups, patients will be treated with FMT totaling three times every 7 days after an antibiotic pretreatment.

Patients randomized to the RYGB- FMT-intervention group will be treated with donor stool from previously obese patients successfully treated with RYGB surgery in terms of maintained weight reduction and improved glucose homeostasis. Patients randomized to Lean-FMT-intervention group will be treated with donor stool from un-operated, metabolically healthy and lean individuals, while patients randomized to the FMT-placebo group will be treated with autologous FMT.

For both allogenic FMT interventions, the donor stool from five different patients successfully treated with RYGB surgery (for RYGB-FMT intervention) and from five un-operated, lean and healthy individuals (for Lean-FMT intervention), respectively, will be anaerobically processed before active study period and stored at - 20° C for analysis and subsequent FMT.

In addition, stool from all 30 obese FMT recipients (FMT-intervention groups and FMT-placebo group) will be collected before the active study period, processed anaerobically and frozen at -80° C. Only stool samples from patients randomized to the FMT-placebo group (n=10) will be used as allogenic transplants.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion criteria for patients

* Age >18 years
* Morbid obesity defined by a BMI ≥ 40 kg/m2
* Prediabetes or diabetes with HbA1C between ≥ 5.7 % OR
* Fasting plasma glucose > 5.6 mmol/l (> 100 mg/dl) (no caloric intake for at least 8 hours) OR
* Random plasma glucose > 11.1 mmol/l (> 200 mg/dl)
* Informed consent

Inclusion criteria for RYGB-FMT intervention donors

* Sustained total weight loss of ≥30% ≥12 months after RYGB surgery
* HbA1c < 6.5% without insulin treatment or oral antidiabetic medication
* Age >18 years
* Informed consent

Inclusion criteria for LEAN-FMT intervention donors

* Normal weight (BMI ≥ 20 to < 25 >18 years
* Informed consent

Exclusion Criteria:

Exclusion criteria for patients

• Non-Compliance

* Insulin dependent diabetes mellitus, treated with GLP-1 agonists or poorly controlled on oral antidiabetic medications (HbA1C > 8%)
* Use of any weight loss medication or participation in a weight loss program
* History of recent body weight change (defined as body weight loss or body weight gain of ≥ 5 kg within the two months preceding study enrolment).
* Use of immunosuppressive medication or immune modulators (glucocorticoids, methotrexate, tacrolimus, cyclosporine, thalidomide, interleukin-10 or -11) within the last three months preceding study enrolment.
* Congenital or acquired immunodeficiencies.
* Anatomical reconstruction of the nutrient passage (i.e. hemicolectomy, resection of small bowel, gastrectomy, sleeve gastrectomy, gastric bypass surgery, biliopancreatic diversion, fundoplication etc) or cholecystectomy.
* Chronic diarrhoea
* History of serious chronic disease including malignancy, rheumatic heart disease, endocarditis, or valvular disease (due to risk of bacteremia)
* Any condition, based on clinical judgment that may make study participation unsafe
* Pregnancy or Breast Feeding

Exclusion criteria for RYGB-FMT intervention donors

* Intake of pre-, pro- or antibiotics within < 3 months before study entry
* Use of immunosuppressive medication or immune modulators (glucocorticoids, methotrexate, tacrolimus, cyclosporine, thalidomide, interleukin-10 or -11) within the last three months preceding study enrolment.
* Congenital or acquired immunodeficiencies.
* Chronic or acute infectious diseases (specified under 6.2.1)
* Drug abuse
* Anatomical reconstruction of the nutrient passage other than surgical RYGB configuration (i.e. hemicolectomy, resection of small bowel, fundoplication, LSG-to-RYGB transformation etc) or cholecystectomy.
* History of recent body weight change (defined as body weight loss or body weight gain of ≥ 5 kg within the two months preceding study enrolment).
* Chronic diarrhoea or steatorrhea or acute gastrointestinal infection within ≤ 3 months before study entry.
* History of serious chronic disease including malignancy, chronic kidney disease (eGFR < 60 ml/min), heart failure (NYHA ≥ III).
* Any further condition, based on clinical judgment that may disqualify the candidate as an appropriate donor.

Exclusion Criteria for Lean-FMT Intervention Donors • History of overweight or obesity in the past (BMI > 25 kg/m2)

• History of recent body weight change (defined as body weight loss or body weight gain of ≥ 5 kg within the two months preceding study enrolment).

• HbA1C > 6.5% or treatment with insulin or oral anti-diabetic medication.

• Use of any weight loss medication or participation in a weight loss program

• Use of immunosuppressive medication or immune modulators (glucocorticoids, methotrexate, tacrolimus, cyclosporine, thalidomide, interleukin-10 or -11) within the last three months preceding study enrolment.

• Congenital or acquired immunodeficiencies.

• Chronic or acute infectious diseases (specified under 6.2.1)

• Drug abuse

• Anatomical reconstruction of the nutrient passage (i.e. hemicolectomy, resection of small bowel, fundoplication etc) or cholecystectomy.

• Chronic diarrhoea or acute gastrointestinal infection within ≤ 3 months before study entry.

• History of serious chronic disease including malignancy, chronic kidney disease (eGFR < 60 ml/min), heart failure (NYHA ≥ III).

• Any further condition, based on clinical judgment that may disqualify the candidate as an appropriate donor.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | after 6 weeks treatment
  Change in insulin sensitivity after FMT compared to baseline as assessed by hyperinsulinemic-euglycemic clamp technique

SECONDARY OUTCOMES:
Insulin sensitivity | after 16/24 weeks treatment
  Change in insulin sensitivity after 16-/24-week treatment compared to baseline as assessed by hyperinsulinemic-euglycemic clamp.
Glucose homeostasis | after 6-/16-/24-week treatment
  Change in glucose homeostasis compared to baseline as assessed by HOMA-IR model, fasting glucose level, and HbA1C value
Body weight | after 6-/16-/24-week treatment
  Change in total body weight, body mass index (BMI) and body composition after 6-/16-/24-week treatment compared to baseline as assessed by Dual-energy X-ray absorptiometry, DXA)
Blood pressure | after 6-/16-/24-week treatment
  Change in blood pressure and antihypertensive medication compared to baseline.
Fasting lipid profile | after 6-/16-/24-week treatment
  Change in fasting lipid profile compared to baseline.
Fasting blood liver enzyme levels | after 6-/16-/24-week treatment
  Change in fasting blood liver enzyme levels and liver fat content (assessed by CAP values with the XL probe) compared to baseline
Dietary intake levels | after 6-/16-/24-week treatment
  Change in dietary intake assessed using MyFitnessPal compared to baseline.
Metabolic inflammation | after 6-/16-/24-week treatment
  Change in metabolic inflammation and endotoxemia as assessed by circulating pro-inflammatory cytokines (TNF-a, IL-6, IL-1ß) and bacterial endotoxins (lipopolysachharide (LPS), LPS-binding protein) compared to baseline
Gut hormones | after 6-/16-/24-week treatment
  Change in postprandial release of gut hormones (PYY, GLP-1, GIP, ghrelin, CCK), insulin and bacterial metabolites (SCFA, Bile acids) before (fasting condition) and during a standardized mixed meal test (MMT) (Fresubin 200ml, 400kcal) compared to baseline
Hunger and Satiety Scores | daily
  Change in Hunger and Satiety Scores assessed via visual analog scales during the MMT
Fecal microbiota composition | after 6-/16-/24-week treatment
  Change in diversity and composition of the fecal microbiota as assessed by 16S rRNA gene profiling compared to baseline
Health-related quality of life | after 6-/16-/24-week treatment
  Change in health-related quality of life and behavior as assessed by established self-report questionnaires compared to baseline measuring: (a) eating behavior including trait food craving (FCQ-T-r), hedonic eating (PFS), restrained eating, overeating, and binge eating (EDE-Q), and emotional eating as well as disinhibition (EI); (b) personality factors such as impulsivity (BIS-15) and reward sensitivity (BIS/BAS); (c) mental and physical health, including depression, anxiety, and substance use (PHQ-D), attention-deficit/hyperactivity disorder (ASRS), and quality of life (EQ-5D). All these questionnaires have established reliability and validity.
Tolerability of repeated FMT | daily
  Safety and tolerability of repeated FMT assessed by review of adverse event diary card

CONTACTS AND LOCATIONS:
Overall Officials: Wiebke K. Fenske, Prof. Dr., Principal Investigator — University Hospital Bergmannsheil Bochum
Locations (1):
- Department of Internal Medicine, Medical University Graz, Graz, Austria

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT06268990/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT06268990/ICF_001.pdf